CLINICAL TRIAL: NCT00001223
Title: Diagnosis and Treatment of Patients With Cystic Fibrosis
Status: Terminated | Type: Observational
Why Stopped: PI left NIH
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 870029; 87-DK-0029
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Cystic Fibrosis; Liver Disease or Abnormalities; Diabetes; Pancreatic Insufficiency (Exocrine and Endocrine)
Keywords: Cystic Fibrosis; Pancreatic Insufficiency; Bronchiectasis; Liver Disease; Natural History
MeSH Terms: conditions — Cystic Fibrosis; Liver Diseases; Congenital Abnormalities; Diabetes Mellitus; Exocrine Pancreatic Insufficiency; Bronchiectasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CF Patients: cystic fibrosis patients
- CF Relatives: relatives of cystic fibrosis patients

SUMMARY:
This is an omnibus protocol for studying patients with cystic fibrosis. The main purpose of the study is to obtain samples and data collected during standard clinical care for future research to expand knowledge of the natural history, clinical manifestations (phenotypes) and the genetic variants (genotypes) of cystic fibrosis.

DETAILED DESCRIPTION:
This is an omnibus protocol for studying patients with cystic fibrosis. The main purpose of the study is to obtain samples and data collected during standard clinical care for future research to expand knowledge of the natural history, clinical manifestations (phenotypes) and the genetic variants (genotypes) of cystic fibrosis.

ELIGIBILITY:
* INCLUSION CRITERIA
* Patients with known or suspected CF and family members of patients with CF.
* >=4 years of age

EXCLUSION CRITERIA

-Concomitant medical, psychiatric or other problems which might complicate interpretation of studies of CF, or for which we are unable to provide adequate care.

Ages: 4 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primarily local population but also any adult patient/relative that moves into the area, either through CF Foundation or relocating for personal reasons.
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 1988-01-01 (Actual); Primary Completion 2026-01-30 (Actual); Study Completion 2026-01-30 (Actual)

PRIMARY OUTCOMES:
To develop a database and collection of samples obtained from patients with CF during their clinical care to allow for future research | end of study
  To develop a collection of samples and a database from patients with cystic fibrosis to be used in future research.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Koh, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
We are open to sharing IPD if requested, but it has not as-to-date been requested from this protocol.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_1987-DK-0029.html